CLINICAL TRIAL: NCT00843882
Title: Randomized Phase III Trial Comparing the Frequency of Major Erythroid Response (MER) to Treatment With Lenalidomide (Revlimid®)) Alone and in Combination With Epoetin Alfa (Procrit®)) in Subjects With Low- or Intermediate-1 Risk MDS and Symptomatic Anemia
Brief Title: Lenalidomide With or Without Epoetin Alfa in Treating Patients With Myelodysplastic Syndrome and Anemia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01173; NCI-2009-01173 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000634119; ECOG-E2905; 09-0095; E2905; E2905 (Other: ECOG-ACRIN Cancer Research Group); E2905 (Other: CTEP); U10CA021115 (NIH); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2021-07-08 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Anemia; Chronic Myelomonocytic Leukemia; De Novo Myelodysplastic Syndrome; Myelodysplastic Syndrome
MeSH Terms: conditions — Anemia; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — Biopsy; Epoetin Alfa; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (lenalidomide) (Active Comparator): Patients receive lenalidomide PO QD on days 1-21. Patients undergo bone marrow biopsy at screening and during follow-up. Patients undergo blood specimen collection on study.
  Interventions: Procedure: Bone Marrow Biopsy; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide
- Arm B (lenalidomide, epoetin alfa) (Experimental): Patients receive lenalidomide PO QD on days 1-21 and epoetin alfa SC once weekly. Patients undergo bone marrow biopsy at screening and during follow-up. Patients undergo blood specimen collection on study.
  Interventions: Procedure: Bone Marrow Biopsy; Biological: Epoetin Alfa; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide

INTERVENTIONS:
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Biological: Epoetin Alfa — Given SC
  Other Names: EPO; Epoetin alfa-epbx; Epogen; Eprex; Procrit; Retacrit
  Arms: Arm B (lenalidomide, epoetin alfa)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid

SUMMARY:
This randomized phase III trial studies lenalidomide to see how well it works with or without epoetin alfa in treating patients with myelodysplastic syndrome and anemia. Lenalidomide may stop the growth of myelodysplastic syndrome by blocking blood flow to the cells. Colony stimulating factors, such as epoetin alfa, may increase the number of immune cells found in bone marrow or peripheral blood. It is not yet known whether lenalidomide is more effective with or without epoetin alfa in treating patients with myelodysplastic syndrome and anemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the rate of major erythroid response (MER) between lenalidomide monotherapy and combined treatment of lenalidomide and epoetin alfa in erythropoietin non-responsive low-/intermediate-1 (Int-1)-risk myelodysplastic syndrome (MDS) patients or erythropoietin treatment naïve patients with low probability of erythropoietin benefit.

SECONDARY OBJECTIVES:

I. To compare the time to MER by treatment assignment. II. To evaluate the duration of MER by treatment assignment. III. To estimate the frequency of MER to salvage combination therapy in patients who fail to experience a MER with lenalidomide monotherapy.

IV. To evaluate and compare the frequency of minor erythroid response by treatment assignment.

V. To investigate the mechanism and target of lenalidomide action in patients with chromosome 5q31.1 deletion.

VI. To evaluate the frequency of cytogenetic response and progression, and the relation between cytogenetic pattern and erythroid response.

VII. To evaluate the frequency of bone marrow response (complete response [CR] + partial response [PR]).

VIII. To evaluate the relationship between erythroid response and laboratory correlates outlined below:

VIIIa. Pretreatment and on study endogenous erythropoietin level (Arm A). VIIIb. To evaluate the effect of CD45 isoform profile on lenalidomide enhancement of erythropoietin-induced STAT5 phosphorylation in CD71^Hi erythroid precursors and the relationship to erythroid response.

VIIIc. To characterize molecular targets relevant to lenalidomide cytotoxicity in del5q31.1 cells.

VIIId. To evaluate the frequency of cryptic chromosome 5q31.1 deletions in patients with non-del5q31.1 MDS by array-based genomic scan, and to determine the relationship to hematologic response.

OUTLINE: Patients are randomized to 1 of 2 treatment arms. Patients with del 5q31.1 karyotype are assigned to Arm A.

ARM A: Patients receive lenalidomide orally (PO) once daily (QD) on days 1-21. Patients undergo bone marrow biopsy at screening and during follow-up. Patients undergo blood specimen collection on study.

ARM B: Patients receive lenalidomide PO QD on days 1-21 and epoetin alfa subcutaneously (SC) once weekly. Patients undergo bone marrow biopsy at screening and during follow-up. Patients undergo blood specimen collection on study.

In both arms, treatment repeats every 28 days for 4 cycles. Patients who achieve a major erythroid response (MER) may continue treatment beyond 4 cycles in the absence of disease progression, disease conversion to acute myeloid leukemia, or unacceptable toxicity. Patients in Arm A who fail to achieve MER or who achieve MER but relapse after 16 weeks of treatment with lenalidomide may crossover and receive treatment in Arm B.

After completion of study treatment, patients are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* NOTE: Results of the bone marrow biopsy and aspirate as well as cytogenetics are mandatory to register subjects onto study, which are indispensable to determine International Prognostic Scoring System (IPSS) category needed for eligibility; please note that it is not necessary to wait for the week 16, week 32, or week bone marrow and cytogenetic results prior to starting the next cycle unless deemed necessary by the treating physician; one example of this exception can include if the subject shows signs of progression, such as increased peripheral blood blast percentage; at that juncture, the treating physician may prefer to await the results prior to starting a new cycle; if a cycle is started, and based on the bone marrow results it is felt by the treating physician that the subject should not continue on treatment, please be sure to note this information on the case report forms at end of treatment
* Patient must have documented diagnosis of MDS lasting at least three months (MDS duration >= 3 months) according to World Health Organization (WHO) criteria or non-proliferative chronic myelomonocytic leukemia (CMML) (white blood cell [WBC] < 12,000/mcL)
* Patient must have International Prognostic Scoring System (IPSS) categories of low- or intermediate-1-risk disease; patients must have IPSS score determined by cytogenetic analysis prior to randomization; patients must have cytogenetic analysis done (to calculate IPSS); if the current bone marrow biopsy is a dry tap, patients with cytogenetic failure and < 10% marrow blasts will be eligible; subjects with cytogenetic failure must have previous cytogenetic results (fluorescence in situ hybridization [FISH] is not a substitute) within the last 6 months post last type of MDS treatment (in this case, not referring to growth factors as type of MDS treatment)
* Must have symptomatic anemia untransfused with hemoglobin < 9.5 g/dL =< 8 weeks prior to randomization or with red blood cells (RBC) transfusion dependence (i.e., >= 2 units/month) confirmed for =< 8 weeks before randomization

  * NOTE: For non-transfusion dependent patients (i.e., receiving < 2 units/4 weeks x 8 weeks pre-study) who receive periodic transfusions, the mean 8 week pre-transfusion hemoglobin should be used to determine protocol eligibility and response reference
  * For non-transfusion dependent patients, a minimum of 2 pre-transfusion or un-transfused hemoglobin values are required
* Applies only for patients without the deletion 5q 31.1; patients must have failed treatment with an erythropoietic growth factor, or have a low probability of response to rhu-erythropoietin; patients with low probability of response to rhu-erythropoietin or prior erythropoietin failures are defined as follows:

  * Prior erythropoietin failure-requires a minimum trial of >= 40,000 units epoetin alfa/week x 8 weeks or equivalent dose of darbepoetin alfa for 8 weeks with failure to achieve transfusion independence in dependent patients or a failure to achieve a >= 2 g rise in hemoglobin sustained for >= 4 weeks in non-transfusion dependent patients
  * Low erythropoietin response profile-rhu-erythropoietin and epoetin alfa-naïve patients receiving >= 2U packed (p)RBC/month for a minimum of 8 weeks, and serum erythropoietin > 500 mU/mL in the 8 weeks prior to randomization for a hemoglobin < 9.5 g/dL
* Patients must be off all non-transfusion therapy for MDS for 28 days prior to initiation of study treatment, including all types of growth factors; patients may receive hydrocortisone prophylactically to prevent transfusion reactions
* Patients must have a serum erythropoietin level documented before randomization and =< 56 days before day 1 of study treatment; NOTE: hemoglobin must be < 9.5 g/dL at time that serum erythropoietin is drawn
* Effective contraception must be used by patients participating in lenalidomide therapy, and all patients must agree to counseling by a trained counselor every 28 days about pregnancy precautions and risks of fetal exposure; females of childbearing potential (FCBP) must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide, during lenalidomide therapy, during dose interruptions, and for at least 28 days following discontinuation of lenalidomide therapy; females of childbearing potential should be referred to a qualified provider of contraceptive methods, if needed; males receiving lenalidomide must agree to use a latex condom during any sexual contact with females of childbearing potential even if they have undergone a successful vasectomy
* Platelet count >= 50,000/mcL (50 x 10^9/L) without platelet transfusion (within 56 days prior to randomization)
* Absolute neutrophil count (ANC) >= 500 cells/mcL (0.5 x 10^9/L); hence ANC must be >= 500/mcL without myeloid growth factor support (within 56 days prior to randomization)
* Serum creatinine =< 1.5 times upper limit of normal (ULN) (within 56 days prior to randomization)
* Serum glutamic oxaloacetic transaminase (SGOT)/aspartate aminotransferase (AST) or serum glutamate pyruvate transaminase (SGPT)/alanine aminotransferase (ALT) =< 2.0 x ULN (within 56 days prior to randomization)
* Serum total bilirubin < 3.0 mg/dL (within 56 days prior to randomization)
* Inclusion criteria for crossover registration from Arm A (lenalidomide alone) to Arm B (lenalidomide and epoetin alfa):
* Patients must have completed 16 weeks of monotherapy with lenalidomide
* Patients must show failure to achieve MER (major erythroid response) or have achieved MER but relapsed on Arm A

Exclusion Criteria:

* Patients must not have documented iron deficiency; all patients must have documented marrow iron stores; if marrow iron stain is not available, the transferrin saturation must be > 20% or a serum ferritin > 100 ng/mL
* Women must not be pregnant or breastfeeding; females of childbearing potential must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days and again within 24 hours prior to starting cycle 1 of lenalidomide; a female of childbearing potential (FCBP) is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months; FCBP must also agree to ongoing pregnancy testing)
* Patients must not have prior therapy with lenalidomide
* Patients must not have a diagnosis of uncontrolled seizure or uncontrolled hypertension
* Patients must not have proliferative (WBC >= 12,000/mcL) chronic myelomonocytic leukemia (CMML); WBC must be < 12,000/mcL
* Patients must not have MDS secondary to treatment with radiotherapy, chemotherapy, and/or immunotherapy for malignant or autoimmune diseases
* Prior thalidomide therapy is allowed, however, patients must not have prior >= grade-3 allergic reactions to thalidomide
* Patients must not have prior history of desquamating rash from thalidomide at time of study entry
* Patients must not have clinically significant anemia resulting from iron, B12 or folate deficiencies, autoimmune or hereditary hemolysis, or gastrointestinal bleeding
* Patients must not have used cytotoxic chemotherapeutic agents or experimental agents (agents that are not commercially available) for the treatment of MDS within 8 weeks of randomization
* Patients must not have prior history of malignancy other than MDS (except basal cell or squamous skin cell carcinoma or carcinoma in situ of the cervix or breast) unless the subject has been confirmed free of disease for >= 3 years
* Patients must not have any serious medical condition or any other unstable medical co-morbidity, or psychiatric illness that will prevent the subject from signing the informed consent form or will place the subject at unacceptable risk if he/she participates in the study
* Patients must not have a history of thrombo-embolic events within 3 years prior to study randomization
* Patients must not have known human immunodeficiency virus (HIV)-1 seropositivity because HIV can be an alternate cause of anemia.
* Patients must not have a known allergic reaction to epoetin alfa (Procrit) or human serum albumin
* Exclusion criteria for crossover registration from Arm A (lenalidomide alone) to Arm B (lenalidomide and epoetin alfa):
* Patients must not have a limiting unresolved grade 3 or greater toxicity from lenalidomide monotherapy or drug intolerance preventing continuation of lenalidomide treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2009-01-29 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2026-10-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Amit K Verma, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (508):
- United States (508):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Saint Helena Hospital, St. Helena, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Leesburg Regional Medical Center, Leesburg, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Augusta University Medical Center, Augusta, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - IU Health Central Indiana Cancer Centers-East, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Premier Oncology Hematology Associates, Merrillville, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - AdventHealth Shawnee Mission, Shawnee Mission, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - King's Daughter's Medical Center, Ashland, Kentucky
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Dana-Farber Cancer Institute at Boston Medical Center - Brighton, Brighton, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Holy Family Hospital, Methuen, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - UP Health System Marquette, Marquette, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Keesler Medical Center, Keesler Air Force Base, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Cheshire Medical Center-Dartmouth-Hitchcock Keene, Keene, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Garnet Health Medical Center, Middletown, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - UNC Rex Healthcare, Raleigh, North Carolina
  - UNC Rex Cancer Center of Wakefield, Raleigh, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Clinton Memorial Hospital/Foster J Boyd Regional Cancer Center, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Butler Memorial Hospital, Butler, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Reading Hospital McGlinn Cancer Institute at Phoenixville, Phoenixville, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - SSM Health Dean Medical Group - South Madison Campus, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] List AF, Sun Z, Verma A, Bennett JM, Komrokji RS, McGraw K, Maciejewski J, Altman JK, Cheema PS, Claxton DF, Luger SM, Mattison RJ, Wassenaar TR, Artz AS, Schiffer CA, Litzow MR, Tallman MS. Lenalidomide-Epoetin Alfa Versus Lenalidomide Monotherapy in Myelodysplastic Syndromes Refractory to Recombinant Erythropoietin. J Clin Oncol. 2021 Mar 20;39(9):1001-1009. doi: 10.1200/JCO.20.01691. Epub 2021 Jan 13. PMID 33439748

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From January 2009 through May 2016, the trial enrolled a total of 247 patients.
Groups:
- Arm A (Lenalidomide; Chromosome 5q31.1 Deletion); Arm A (Lenalidomide; Randomization): Patients receive lenalidomide PO QD on days 1-21.
- Arm B (Lenalidomide + Epoetin Alfa; Randomization): Patients receive lenalidomide PO QD on days 1-21 and epoetin alfa SC once weekly.
Period: Step 1
Arm/Group | Arm A (Lenalidomide; Chromosome 5q31.1 Deletion) | Arm A (Lenalidomide; Randomization) | Arm B (Lenalidomide + Epoetin Alfa; Randomization)
Started | 38 | 103 | 106
Treated Patients | 36 | 103 | 106
Evaluable Patients Included in Primary Analysis | 0 | 96 | 99
Patients With Cytogenetic Response Data Available | 0 | 55 | 51
Completed | 6 | 48 | 41
Not Completed | 32 | 55 | 65
Not completed — Lack of Efficacy | 14 | 10 | 21
Not completed — Adverse Event | 8 | 17 | 20
Not completed — Death | 1 | 2 | 4
Not completed — Withdrawal by Subject | 6 | 12 | 9
Not completed — Physician Decision | 0 | 5 | 1
Not completed — Patient and physician's decision | 0 | 0 | 1
Not completed — Other complicating disease | 1 | 3 | 4
Not completed — Alternative therapy | 0 | 1 | 1
Not completed — Patient switched treatment early due to DSMC announcement | 0 | 4 | 0
Not completed — Off treatment reason unknown | 0 | 1 | 4
Not completed — Never started treatment | 2 | 0 | 0
Period: Step 2 (Cross-over to Arm B)
Arm/Group | Arm A (Lenalidomide; Chromosome 5q31.1 Deletion) | Arm A (Lenalidomide; Randomization) | Arm B (Lenalidomide + Epoetin Alfa; Randomization)
Started | 7 (All patients in Arm A that did not achieve major erythroid response (MER) were offered to receive combined treatment in Step 2.) | 46 (All patients in Arm A that did not achieve major erythroid response (MER) were offered to receive combined treatment in Step 2.) | 0 (Only patients in Arm A that did not achieve major erythroid response (MER) were offered to receive combined treatment in Step 2.)
Evaluable Patients Included in Primary Analysis | 7 | 37 | 0
Completed | 3 | 20 | 0
Not Completed | 4 | 26 | 0
Not completed — Lack of Efficacy | 1 | 9 | 0
Not completed — Adverse Event | 0 | 6 | 0
Not completed — Death | 0 | 3 | 0
Not completed — Withdrawal by Subject | 2 | 5 | 0
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Alternative treatment | 0 | 1 | 0
Not completed — Prolonged wound healing | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All patients enrolled are included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Lenalidomide; Chromosome 5q31.1 Deletion) | Arm A (Lenalidomide; Randomization) | Arm B (Lenalidomide + Epoetin Alfa; Randomization) | Total
Number analyzed (Participants) | 38 | 103 | 106 | 247
Age, Continuous [Median (Full Range); unit: years] | 77 [62 to 88] | 74 [49 to 89] | 73 [47 to 92] | 74 [47 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 33 | 28 | 87
  Male | 12 | 70 | 78 | 160
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 5
  Not Hispanic or Latino | 34 | 96 | 97 | 227
  Unknown or Not Reported | 2 | 5 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 3 | 4
  White | 35 | 97 | 96 | 228
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Major Erythroid Response (MER)
Description: Major erythroid response is defined as transfusion-independence for ≥ 8 consecutive weeks for patients who were red blood cell transfusion-dependent at baseline AND a ≥ 1 g/dL hemoglobin rise compared to mean pre-transfusion baseline value; or a > 2 g/dL rise in hemoglobin without transfusion for non-transfusion dependent patients.
Time Frame: Assessed after completion of 16 weeks of treatment
Population: Evaluable patients randomized to either arm A or arm B
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Lenalidomide; Randomization) | Arm B (Lenalidomide + Epoetin Alfa; Randomization)
Number analyzed (Participants) | 96 | 99
proportion of participants | 0.115 [0.066 to 0.183] | 0.283 [0.209 to 0.367]
Statistical Analysis 1: Comparison: Arm A (Lenalidomide; Randomization) vs Arm B (Lenalidomide + Epoetin Alfa; Randomization); Test type: Superiority; p = 0.004, Fisher Exact

2. Secondary Outcome: Time to Major Erythroid Response (MER)
Description: Time to major erythroid response (MER) is defined in responders as the time from randomization to the documented date of MER.
  For transfusion independent patients, the date of MER is the first date of the elevation in hemoglobin level of more than 2 g/dL that has been sustained for at least 8 weeks. For transfusion dependent patients, the date of MER is the beginning date of the time interval of transfusion independence that has been sustained for at least eight weeks.
Time Frame: Assessed every cycle during treatment and then 3 and 6 months after last protocol treatment
Population: Only evaluable patients who achieved MER among randomized patients were included in this analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A (Lenalidomide; Randomization) | Arm B (Lenalidomide + Epoetin Alfa; Randomization)
Number analyzed (Participants) | 11 | 28
months | 3.6 [2.1 to 5.5] | 3.7 [1.0 to 10.6]

3. Secondary Outcome: Duration of Major Erythroid Response (MER)
Description: Duration of major erythroid response (MER) is defined as the time interval between the documented date of MER and the earliest date of resumption of red blood cell transfusions ≥ 2 units in an 8-week period, a reduction in hemoglobin concentration ≥ 2 g/dL in the absence of acute infection, gastrointestinal bleeding and hemolysis, or death.
Time Frame: Assessed every cycle during treatment and then 3 and 6 months after last protocol treatment
Population: Only evaluable patients who achieved MER among randomized patients were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Lenalidomide; Randomization) | Arm B (Lenalidomide + Epoetin Alfa; Randomization)
Number analyzed (Participants) | 11 | 28
months | 13 [2.1 to 75] | 23.8 [8.5 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

4. Secondary Outcome: Proportion of Patients With Major Erythroid Response (MER) to Salvage Combination Therapy
Description: as for outcome 1
Time Frame: Assessed after completion of 16 weeks of treatment
Population: Evaluable patients who fail to experience a MER with lenalidomide monotherapy and receive salvage combination therapy (crossover from arm A to arm B)
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Arm B (Lenalidomide + Epoetin Alfa; Crossover): Patients receive lenalidomide PO QD on days 1-21 and epoetin alfa SC once weekly.
Arm/Group | Arm B (Lenalidomide + Epoetin Alfa; Crossover)
Number analyzed (Participants) | 44
proportion of participants | 0.25 [0.13 to 0.40]

5. Secondary Outcome: Proportion of Patients With Minor Erythroid Response
Description: The definition of minor erythroid response: the mean hemoglobin is sustained 1.0 to 2.0 g/dL above the baseline value for a minimum of 8 weeks; or a 50% or greater decrease in 8-week red blood cell transfusion requirements compared to baseline.
Time Frame: Assessed every cycle during treatment and after completion of 16 weeks of treatment
Population: Evaluable patients randomized to either arm A or arm B
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Lenalidomide; Randomization) | Arm B (Lenalidomide + Epoetin Alfa; Randomization)
Number analyzed (Participants) | 96 | 99
proportion of participants | 0.208 [0.142 to 0.288] | 0.182 [0.121 to 0.258]

6. Secondary Outcome: Proportion of Patients With Major Erythroid Response (MER) Among Those With Chromosome 5q31.1 Deletion
Description: as for outcome 1
Time Frame: Assessed after completion of 16 weeks of treatment
Population: All patients with chromosome 5q31.1 deletion in arm A
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Lenalidomide; Chromosome 5q31.1 Deletion)
Number analyzed (Participants) | 38
proportion of participants | 0.632 [0.46 to 0.782]

7. Secondary Outcome: Proportion of Patients With Bone Marrow Response
Description: Bone marrow response includes complete remission (CR) and partial remission (PR).
  Complete remission (CR): Bone marrow showing < 5% myeloblasts with normal maturation of all cell lines, with no evidence for dysplasia. When erythroid precursors constitute < 50% of bone marrow nucleated cells, the percent of blasts is based on all nucleated cells; when there are ≥ 50% erythroid cells, the percent blasts should be based on the non-erythroid cells.
  Partial remission (PR): All of the CR criteria (if abnormal prior to treatment), except blasts decreased by 50% over pre-treatment, or a less advanced Myelodysplastic Syndromes (MDS) World Health Organization (WHO) classification than pretreatment. Cellularity and morphology are not relevant.
Time Frame: Assessed at 16 weeks
Population: Evaluable patients randomized to either arm A or arm B
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Lenalidomide; Randomization) | Arm B (Lenalidomide + Epoetin Alfa; Randomization)
Number analyzed (Participants) | 96 | 99
proportion of participants | 0.01 [0.0006 to 0.049] | 0.03 [0.008 to 0.077]

8. Secondary Outcome: Proportion of Patients With Cytogenetic Response
Description: Evaluation of cytogenetic response requires 20 analyzable metaphases when using conventional techniques. Analysis of data will require 20 metaphases before and after treatment, which must be done on bone marrow only (peripheral blood is not a substitute). Fluorescent in situ hybridization (FISH) may be used as a supplement to follow a specifically defined cytogenetic abnormality, but it is not a substitute for conventional cytogenetic studies. Cytogenetic response is defined as follows: Complete response: Restoration of a normal karyotype in patients with a documented pre-existing clonal (>2 metaphases abnormal) chromosome abnormalities.
  Partial response: > 50% reduction in the percentage of bone marrow metaphases with only clonal abnormality.
Time Frame: Assessed at baseline and after completion of 16 weeks of treatment
Population: Evaluable patients randomized to either arm A or arm B who had cytogenetic response data
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Lenalidomide; Randomization) | Arm B (Lenalidomide + Epoetin Alfa; Randomization)
Number analyzed (Participants) | 55 | 51
proportion of participants | 0.07 [0.02 to 0.18] | 0.10 [0.03 to 0.21]

9. Secondary Outcome: Association Between Major Erythroid Response and Cytogenetic Response
Description: Major erythroid response is defined as transfusion-independence for ≥ 8 consecutive weeks for patients who were red blood cell transfusion-dependent at baseline AND a ≥ 1 g/dL hemoglobin rise compared to mean pre-transfusion baseline value; or a > 2 g/dL rise in hemoglobin without transfusion for non-transfusion dependent patients.
  Evaluation of cytogenetic response requires 20 analyzable metaphases before and after treatment, which must be done on bone marrow only. Fluorescent in situ hybridization (FISH) may be used as a supplement to follow a specifically defined cytogenetic abnormality, but it is not a substitute for conventional cytogenetic studies. Cytogenetic response is defined as follows:
  Complete response: Restoration of a normal karyotype in patients with a documented pre-existing clonal (>2 metaphases abnormal) chromosome abnormalities.
  Partial response: > 50% reduction in the percentage of bone marrow metaphases with only clonal abnormality.
Time Frame: Assessed at baseline and after completion of 16 weeks of treatment
Population: Evaluable patients in both arms A and B who had both major erythroid response data and cytogenetic response data
Measure: Count of Participants; unit: Participants
Groups:
- Major Erythroid Response: Patients with major erythroid response
- No Major Erythroid Response: Patients without major erythroid response
Arm/Group | Major Erythroid Response | No Major Erythroid Response
Number analyzed (Participants) | 23 | 83
Participants
  Cytogenetic response | 4 | 5
  No cytogenetic response | 19 | 78

10. Secondary Outcome: Pretreatment Endogenous Erythropoietin Level
Description: Pretreatment endogenous erythropoietin level was assessed at baseline. The association between pretreatment endogenous erythropoietin level and major erythroid response was evaluated among patients who received lenalidomide alone.
  Major erythroid response is defined as transfusion-independence for ≥ 8 consecutive weeks for patients who were red blood cell transfusion-dependent at baseline AND a ≥ 1 g/dL hemoglobin rise compared to mean pre-transfusion baseline value; or a > 2 g/dL rise in hemoglobin without transfusion for non-transfusion dependent patients.
Time Frame: Assessed at baseline and after completion of 16 weeks of treatment
Population: All patients randomized to arm A and all patients with 5q31.1 deletion that received lenalidomide alone
Measure: Median (Full Range); unit: mU/mL
Groups:
- Arm A Patients With Major Erythroid Response; Arm A Patients Without Major Erythroid Response: Patients receive lenalidomide PO QD on days 1-21 and achieve major erythroid response.
Arm/Group | Arm A Patients With Major Erythroid Response | Arm A Patients Without Major Erythroid Response
Number analyzed (Participants) | 36 | 105
mU/mL | 514.5 [82 to 3405] | 150 [11 to 3048]
Statistical Analysis 1: Comparison: Arm A Patients With Major Erythroid Response vs Arm A Patients Without Major Erythroid Response; Test type: Superiority; p = 0.0002, Wilcoxon (Mann-Whitney)

11. Other Pre Specified Outcome: The Association Between CD45 Isoform Profile and ex Vivo Augmentation of STAT5 Phosphorylation by Lenalidomide
Description: To evaluate the effect of CD45 isoform profile on lenalidomide enhancement of erythropoietin-induced STAT5 phosphorylation in CD71Hi erythroid precursors and the relationship to erythroid response.
Time Frame: Assessed at baseline and after completion of 16 weeks of treatment
Reporting Status: Not Posted

12. Other Pre Specified Outcome: RNA and Protein Expression Level of Cdc25C, PP2A and Their Phosphatase Substrates, Cdc2phospho-Tyr15 and Cdc25Cphospho-Ser216
Description: To characterize molecular targets relevant to lenalidomide cytotoxicity in del5q31.1 cells.
Time Frame: Assessed at baseline and after completion of 16 weeks of treatment
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Proportion of Patients With Cryptic Chromosome 5q31.1 Deletions
Description: To evaluate the frequency of cryptic chromosome 5q31.1 deletions in patients with non-del5q31.1 MDS by array based genomic scan, and to determine the relationship to hematologic response.
Time Frame: Assessed at baseline and after completion of 16 weeks of treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment
Description: Adverse events were assessed among patients who started protocol treatment. All-cause mortality was assessed among all registered patients.
Groups:
- Arm A (Step 1; Regardless of Chromosome 5q31.1 Status): Patients receive lenalidomide PO QD on days 1-21.
- Arm B (Step 1 Randomization; Lenalidomide + Epoetin Alfa); Arm B (Step 2 Cross-over; Lenalidomide + Epoetin Alfa): Patients receive lenalidomide PO QD on days 1-21 and epoetin alfa SC once weekly.
Arm/Group | Arm A (Step 1; Regardless of Chromosome 5q31.1 Status) | Arm B (Step 1 Randomization; Lenalidomide + Epoetin Alfa) | Arm B (Step 2 Cross-over; Lenalidomide + Epoetin Alfa)
All-Cause Mortality (participants affected / at risk) | 29/141 | 29/106 | 0/53
Serious Adverse Events (participants affected / at risk) | 123/139 | 98/106 | 49/53
Other Adverse Events (participants affected / at risk) | 137/139 | 105/106 | 52/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Step 1; Regardless of Chromosome 5q31.1 Status) (N=139) | Arm B (Step 1 Randomization; Lenalidomide + Epoetin Alfa) (N=106) | Arm B (Step 2 Cross-over; Lenalidomide + Epoetin Alfa) (N=53)
Anemia (Blood and lymphatic system disorders) | 80 | 65 | 30
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 4 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 1 | 0
Heart failure (Cardiac disorders) | 1 | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 1 | 0
Edema limbs (General disorders) | 1 | 1 | 1
Fatigue (General disorders) | 4 | 8 | 2
Fever (General disorders) | 0 | 2 | 0
Multi-organ failure (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 3 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 3 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Anaphylaxis (Immune system disorders) | 0 | 1 | 0
Immune system disorders - Other, specify (Immune system disorders) | 0 | 1 | 0
Bronchial infection (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 2 | 2 | 0
Sepsis (Infections and infestations) | 1 | 2 | 0
Soft tissue infection (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1
Infections and infestations - Other (Infections and infestations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 0
Creatinine increased (Investigations) | 3 | 5 | 1
Hemoglobin increased (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 4 | 5 | 2
Neutrophil count decreased (Investigations) | 92 | 69 | 39
Platelet count decreased (Investigations) | 45 | 28 | 9
Weight gain (Investigations) | 0 | 1 | 0
White blood cell decreased (Investigations) | 50 | 36 | 24
Investigations - Other, specify (Investigations) | 0 | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Iron overload (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Leukemia secondary to oncology chemo (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasms - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Optic nerve disorder (Eye disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory thoracic mediastinal - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Step 1; Regardless of Chromosome 5q31.1 Status) (N=139) | Arm B (Step 1 Randomization; Lenalidomide + Epoetin Alfa) (N=106) | Arm B (Step 2 Cross-over; Lenalidomide + Epoetin Alfa) (N=53)
Anemia (Blood and lymphatic system disorders) | 108 | 92 | 43
Fatigue (General disorders) | 11 | 10 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 | 5 | 0
Diarrhea (Gastrointestinal disorders) | 7 | 3 | 0
Creatinine increased (Investigations) | 62 | 50 | 15
Neutrophil count decreased (Investigations) | 99 | 73 | 43
Platelet count decreased (Investigations) | 108 | 77 | 38
White blood cell decreased (Investigations) | 114 | 91 | 47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT00843882/Prot_SAP_000.pdf